CLINICAL TRIAL: NCT04391153
Title: Fluorescent in Situ Hybridization in Diagnosis of Biliary Stricture: A Feasibility Study
Brief Title: FISH in Diagnosis of Biliary Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Vincent Zoundjiekpon, principal investigator, University Hospital Olomouc
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UHO003
Record Dates: First submitted 2020-05-10; First posted 2020-05-18 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Biliary Stricture
Keywords: suspected malignant biliary stricture; fluorescence in situ hybridization; endoscopic retrograde cholangiopancreatography; brushing; forceps biopsy; endosonography/ EUS-FNA
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional samplig (Active Comparator): Patients with biliary strictures udergo ERCP or EUS. Tissue specimens obtained via either of brush cytology, forceps biopsy or fine needle aspiration during ERCP or endosonography (EUS) were examined by routine cytology or histology methods.
  Gold standard for final diagnosis is the histology from surgical resection. In patients without surgery, a follow up of 12 months will be considered adequate to exclude or confirm malignant etiology.
  Interventions: Procedure: ERCP with tissue sampling
- Fluorescence in situ Hybridization (FISH) (Active Comparator): Tissue specimens obtained via either of brush cytology, forceps biopsy or fine needle aspiration during ERCP or endosonography (EUS) were examined by routine cytology or histology methods. In addition, FISH inlcuding fluorescence-based polynucleotide probes targeting chromosomes 3, 7, 17 and locus 9p21 was performed. Gold standard for final diagnosis is the histology from surgical resection. In patients without surgery, a follow up of 12 months will be considered adequate to exclude or confirm malignant etiology.
  Interventions: Procedure: ERCP with tissue sampling

INTERVENTIONS:
Procedure: ERCP with tissue sampling — Patients with biliary strictures undergo ERCP o EUS. Tissue specimens obtained via either of brush cytology, forceps biopsy or fine needle aspiration during ERCP or endosonography (EUS) were examined by routine cytology or histology methods. In addition, FISH inlcuding fluorescence-based polynucleotide probes targeting chromosomes 3, 7, 17 and locus 9p21 was performed. Gold standard for final diagnosis is the histology from surgical resection. In patients without surgery, a follow up of 12 months will be considered adequate to exclude or confirm malignant etiology.

SUMMARY:
The management of biliary strictures depends on their correct pre-operative evaluation which remains challenging. Despite the emerging multitudes of new diagnostic opportunities- modalities we have today, there is still a large number of biliary stenosis misdiagnosed with a profound negative impact on the patients´ outcome. The study aims to proove the feasibility and to evaluate the impact of Fluorescent In Situ Hybridization (FISH) on the tissue diagnostic of biliary strictures.

DETAILED DESCRIPTION:
The management of biliary strictures depends on their correct pre-operative evaluation which remains challenging. Biliary strictures have various etiologies (traumatic, inflammatory, tumoral, ischemic etc), which are necessarily needed to be known for the correct therapeutic approach. Despite the emerging multitudes of new diagnostic opportunities, there is still a large number of biliary stenosis misdiagnosed with a profound negative impact on the patients´ outcome. The dilemma that exists is how to balance the risk of missing the chance of curative surgery for some malignancy and preventing some patients from unnecessary surgery for benign etiologies and not to waste time. Different conventionnal sampling methods (as Brush-cytology, forceps biopsies during ERCP, endoscopic guided fine needle aspiration-EUS-FNA) have relatively low sensitivity. In such cases, the peroral cholangioscopy proves diagnostic accuracy of 90 %. This method remains expert dependent, costly and may be result in complications of cholangitis in 3-5 % of cases. Techniques or others methods less complicated and improving the preoperative diagnosis of biliary strictures are needed. Fluorescent in Situ Hybridization (FISH) was shown to improve the diagnostic yield of routine cytology.

This study will proove the feasebility and the clinical place of FISH in the diagnostic of biliary strictures and evaluate the impact of FISH on management of patients with biliary strictures.

FISH (Fluorecent In Situ Hybridization) is a molecular cytogenetic method, which enables the detection of fluorescently- labeled DNA/RNA or oligonucleotide probes hybridized to metaphase/ interphase. It uses probes to bind to specific DNA/RNA sequences. This enables the detection of aneuploidy for chromosomes 3, 7, 17 and loss of the 9p21 in patients with suspected malignant biliary strictures.

Different methods were used to take samples from the site of the stenosis. Brush-cytology and endocanal forceps biopsies during ERCP and FNA (fine needle aspiration) during EUS (endosonography). These sampling techniques have relatively low specificity and sensitivity. Reason why we will combine FISH with the sampling methods to maximize our chance to early determine the etiology of stenosis and avoid wasting time and unnecessary cholangioscopy. In this study, the positivity of FISH for Chromosomes 3,7,17 is defined by a presence of polysomy of these chromosomes and the positivity of FISH for Chromosomal region defined by a presence of heterozygous delection or homozygous delection for 9p21. Polysomy is defined by a gain of 2 or more chromosomes in 4 cells. For the chromosomal region, the delection or loss of 9p21 must be observed in 12 cells.

Methods:

* Tissue specimens obtained via either brush cytology, forceps biopsy or fine needle aspiration during ERCP or endosonography (EUS) were examined by routine cytology or histology (RC) methods.
* In addition, FISH using fluorescent-based polynucleotide probes targeting chromosomes 3, 7, 17 and locus 9p21 was performed (ZytoVysion®).

Success (positivity) is defined by the presence of polysomy for chromosomes 3, 7, 17 and/or the presence of delection or loss of the chromosomal region 9p21 in patients with suspected malignant biliary strictures.

Gold standard for final diagnosis should be the histology from surgery resection. In patients without surgery, a follow up of 12 months will be considered adequate to exclude or confirm malignant etiology of the stritures.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected malignant biliary stricture
2. Localization: Extrahepatic biliary duct
3. Patient´s consent with a diagnostic procedure
4. Age : 18 years or more

Exclusion Criteria:

1. Intrahepatic biliary strictures
2. Duodenal stenosis (endoscopically)
3. Age : < 18 years
4. Coagulopathy : (INR >1,5, Platelets < 100)
5. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-05-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-19 (Estimated)

PRIMARY OUTCOMES:
Proove the feasebility and the clinical place of FISH in the diagnostic of biliary strictures | 1- 7 days
  The the sensitivity (%) and specificity (%) of ERCP/ EUS with conventional tissue sampling - Brushing, forceps biopsy/EUS-FNA and ERCP/EUS with conventional tissue sampling completed with FISH in patients with suspected malignant stricture of the common bile duct are evaluated. Success (positivity) is defined by the presence of benign or malignant cells, adequate to make the final tissue diagnosis. Based on the previous studies and the experiences of our endoscopists and pathologist, we can expect the diagnostic yield with FISH will be increased of 20-30% in the study population (the samples size 96).

SECONDARY OUTCOMES:
evaluate the impact of FISH on management of patients with biliary stricture. | 3-6 months
  The proportion of patients (%) who will miss the chance of curative surgery for some malignancy and the proportion of patients (%) who will not have unnecessary surgery for benign etiologies are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Zoundjiekpon, MD, Principal Investigator — 2nd Department of Internal Medicine, University Hospital Olomouc, Czech Republic
Locations (1):
- 2nd Department of Internal Medicine, University Hospital and Palacký University,, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No